CLINICAL TRIAL: NCT01750138
Title: Can Preoperative Oral Glutamine Facilitate Earlier Return of Gut Function in Patients Undergoing Colorectal Surgery. A Prospective Randomized Trial.
Brief Title: SNE1725: Can Oral Glutamine Facilitate Early Return of Gut Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scarborough General Hospital (Other)
Responsible Party: Principal Investigator, Syed Irfan Kabir, Research Fellow, Scarborough General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SNE1725
Record Dates: First submitted 2012-12-11; First posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Gut Function
MeSH Terms: interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glutamine (Experimental): Glutamine powder given preoperatively for five days
  Interventions: Drug: Glutamine
- Placebo (Active Comparator): dextrose powder for 5 days pre-operatively
  Interventions: Drug: Dextrose powder

INTERVENTIONS:
Drug: Glutamine
  Arms: Glutamine
Drug: Dextrose powder
  Arms: Placebo

SUMMARY:
The gastrointestinal tract has many functions; it provides nutrition, produces hormones, performs a barrier function, maintains a stable gastrointestinal micro flora and plays an important role in the inflammatory process as it is the largest producer of cytokines (proteins associated with inflammation). This gut function is impaired after colorectal (bowel) surgery. There is evidence to suggest that impaired gut function is associated with increased complications. Hence if gut function is preserved, it should equate with better outcomes. As a result, there has been increasing interest in treatments called Gut Specific Nutrients (GSN), which specifically target gut function. Most notable of them is Glutamine, a conditionally essential amino acid and preferred fuel source for intestinal cells. Research has shown that glutamine promotes cell growth, increases clearance of harmful organisms from the blood, and reduces the surgical stress response. In other words, glutamine has a favourable influence on gut function.

Recent studies from our unit using intravenous glutamine in critically ill patients have shown an early return of gut function, which in turn is associated with attenuation of the inflammatory response and improved outcomes. It is not known whether oral glutamine is associated with a similar outcome. A recent pilot study at our unit suggests an association between oral glutamine and early return of gut function. The aim of this research is to determine if giving oral glutamine results in an early return of gut function and whether this is associated with an attenuation of the systemic inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing elective colorectal surgery (both open or keyhole) will be eligible for the study.

Exclusion Criteria:

* Allergy to glutamine/placebo
* Failure to obtain informed consent.
* Patients with existing infections.
* Pregnant women and children under the age of 18 years will be excluded from the study.
* Patients on antibiotics in the previous 2 weeks.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Gut function | post op

CONTACTS AND LOCATIONS:
Overall Officials: syed irfan kabir, MBBS, MSc, Principal Investigator — Scarborough General Hospital
Locations (1):
- Scarborough District Hospital, Scarborough, North Yorkshire, United Kingdom